CLINICAL TRIAL: NCT00522951
Title: Multi-center, Randomized, Controlled, Single-blind, Intra-individual Comparisons of 2 Dose of Gadobutrol 1.0 Molar and Gadoteridol (ProHance) Crossover Studies With Corresponding Blinded Image Evaluation Following Multiple Injections of 0.1 mmol/kg bw of Gadobutrol and Gadoteridol in Patients With Known or Suspected Brain Metastasis
Brief Title: SH L 562BB Phase II/III Dose Justification and Gadoteridol-controlled Comparative Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 91569; 310864 (Other: Company internal)
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-07

CONDITIONS: Brain Metastases
Keywords: MRI; Brain Metastasis; Gadolinium; Imaging; Diagnostic Agent
MeSH Terms: conditions — Brain Neoplasms | interventions — gadobutrol; gadoteridol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gadobutrol 0.1 mmol/kg bw (Experimental): Participants received first injection (intravenous [i.v.]) of gadobutrol 0.1 mmol/kg body weight (bw), corresponding to a dose of 0.1 mmol/kg bw
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)
- Gadobutrol 0.2 mmol/kg bw (Experimental): Participants received second injection (i.v.) of gadobutrol 0.1 mmol/kg bw, corresponding to a total dose of 0.2 mmol/kg bw. The interval of two bolus injections is 13-15 min
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)
- Gadoteridol (ProHance) (Experimental): Participants received two injections (i.v.) of gadoteridol 0.1 mmol/kg bw, corresponding to a total dose of 0.2 mmol/kg bw. The interval of two bolus injections is 13-15 min
  Interventions: Drug: ProHance

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — Gadobutrol enhanced MRI (first injection of gadobutrol 0.1 mmol/kg bw, corresponding to a dose of 0.1 mmol/kg bw)
  Arms: Gadobutrol 0.1 mmol/kg bw
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — Gadobutrol enhanced MRI (second injection of gadobutrol 0.1 mmol/kg bw, corresponding to a total dose of 0.2 mmol/kg bw)
  Arms: Gadobutrol 0.2 mmol/kg bw
Drug: ProHance — ProHance enhanced MRI (two injections of gadoteridol 0.1 mmol/kg bw, corresponding to a total dose of 0.2 mmol/kg bw)
  Arms: Gadoteridol (ProHance)

SUMMARY:
This study is conducted to compare the contrast effect and safety of SH L562BB with ProHance, which has already been approved as a pharmaceutical product of similar indication.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients at least 20 years of age
* Patients with diagnosed primary cancer
* Patients with metastatic lesions by CT/MRI

Exclusion Criteria:

* Patients who have contraindication to the MRI examinations
* Patients who have severe renal disorder
* Patients in extremely serious general condition

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (18):
- Japan (18):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Kitakyushu, Fukuoka
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Habikino, Osaka
  - Sayama, Osaka
  - Hamamatsu, Shizuoka
  - Sunto, Shizuoka
  - Bunkyo-ku, Tokyo
  - Chuo-ku, Tokyo
  - Mitaka, Tokyo
  - Shinagawa-ku, Tokyo
  - Yonago, Tottori
  - Fukuoka
  - Osaka

REFERENCES:
- [Result] Katakami N, Inaba Y, Sugata S, Tsurusaki M, Itoh T, Machida T, Tanaka H, Nakayama T, Morikawa T, Breuer J, Aitoku Y. Magnetic resonance evaluation of brain metastases from systemic malignances with two doses of gadobutrol 1.0 m compared with gadoteridol: a multicenter, phase ii/iii study in patients with known or suspected brain metastases. Invest Radiol. 2011 Jul;46(7):411-8. doi: 10.1097/RLI.0b013e3182145a6c. PMID 21467949

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 175 participants were enrolled into the study. 10 were withdrawn from the study before entering Study Period 1. Safety Analysis Set included 164 participants; gadobutrol=161, ProHance=162. Per Protocol Set (PPS) included 151 participants.
Groups:
- Gadobutrol Then Gadoteridol: Participants who received two injections of gadobutrol 0.1 mmol/kg body weight (bw) in Period 1, and two injections of gadoteridol 0.1 mmol/kg bw in Period 2
- Gadoteridol Then Gadobutrol: Participants who received two injections of gadoteridol 0.1 mmol/kg body weight (bw) in Period 1, and two injections of gadobutrol 0.1 mmol/kg bw in Period 2
Period: Period 1
Arm/Group | Gadobutrol Then Gadoteridol | Gadoteridol Then Gadobutrol
Started | 86 | 79
Received Treatment | 86 | 78
Completed | 86 | 78
Not Completed | 0 | 1
Not completed — body motion | 0 | 1
Period: Washout Period
Arm/Group | Gadobutrol Then Gadoteridol | Gadoteridol Then Gadobutrol
Started | 86 | 78
Completed | 86 | 76
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Death | 0 | 1
Period: Period 2
Arm/Group | Gadobutrol Then Gadoteridol | Gadoteridol Then Gadobutrol
Started | 86 | 76
Subjects Received Treatment | 84 | 75
Completed | 84 | 75
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — residual contrast medium | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: includes all participants received treatment
Arm/Group | Entire Study Population
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 90
Height [Mean (Standard Deviation); unit: cm] | 160.9 (8.7)
Body weight [Mean (Standard Deviation); unit: kg] | 56.7 (12.2)
Primary focus [Number; unit: participants]
  Lung cancer | 123
  Breast cancer | 20
  Others | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Lesions Detected by Blinded Readers (BR) and Investigator
Description: Number of metastatic lesions (unenhanced and enhanced) per participant detected on postcontrast Magnetic resonance (MR) images by averaged blinded reader and investigator
Time Frame: one day
Population: Participants without a major protocol deviation or conditions that could affect his or her efficacy evaluation (Per Protocol Set), with valid data for this Outcome Measure.
Measure: Mean (Standard Deviation); unit: lesions
Groups:
- Gadoteridol (ProHance) 0.2mmol/kg bw: Participants received two injections (i.v.) of gadoteridol 0.1 mmol/kg bw, corresponding to a total dose of 0.2 mmol/kg bw. The interval of two bolus injections is 13-15 min
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 151 | 151 | 151
lesions
  averaged blinded reader | 6.28 (8.31) | 6.92 (8.69) | 6.87 (8.65)
  investigator | 6.36 (8.26) | 6.87 (8.49) | 6.66 (8.41)
Statistical Analysis 1: Comparison: Gadobutrol 0.1 mmol/kg bw vs Gadoteridol (ProHance) 0.2mmol/kg bw; H01: μG1 - μPr ≤ -1; Test type: Non-Inferiority or Equivalence — non-inferiority margin = -1; Mean Difference (Final Values) = -0.58, 95% CI [-0.87 to -0.29] — Averaged blinded reader (primary analysis)
Statistical Analysis 2: Comparison: Gadobutrol 0.2 mmol/kg bw vs Gadoteridol (ProHance) 0.2mmol/kg bw; H02: μG2 - μPr ≤ -1; Test type: Non-Inferiority or Equivalence — non-inferiority margin = -1; Mean Difference (Final Values) = 0.06, 95% CI [-0.23 to 0.36] — Averaged blinded reader (primary analysis)
Statistical Analysis 3: Comparison: Gadobutrol 0.1 mmol/kg bw vs Gadoteridol (ProHance) 0.2mmol/kg bw; H01: μG1 - μPr ≤ -1; Test type: Non-Inferiority or Equivalence — non-inferiority margin = -1; Mean Difference (Final Values) = -0.3, 95% CI [-0.5 to -0.1] — Investigator (secondary analysis)
Statistical Analysis 4: Comparison: Gadobutrol 0.2 mmol/kg bw vs Gadoteridol (ProHance) 0.2mmol/kg bw; H02: μG2 - μPr ≤ -1; Test type: Non-Inferiority or Equivalence — non-inferiority margin = -1; Mean Difference (Final Values) = 0.21, 95% CI [0.02 to 0.41] — Investigator (secondary analysis)

2. Secondary Outcome: Score of Visibility Assessment - Degree of Lesion Contrast Enhancement by Blinded Reader
Description: Degree of contrast enhancement for each lesion on postcontrast MR images using the 4-point scale by averaged blinded reader (Score 1=No, 2=Moderate, 3=Good, 4=Excellent)
Time Frame: one day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 143 | 148 | 149
scores on a scale | 3.44 (0.42) | 3.54 (0.44) | 3.51 (0.49)

3. Secondary Outcome: Score of Visibility Assessment - Degree of Lesion Contrast Enhancement by Investigator
Description: Degree of contrast enhancement for each lesion on postcontrast MR images using the 4-point scale by investigator (Score 1=No, 2=Moderate, 3=Good, 4=Excellent)
Time Frame: one day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 143 | 143 | 144
scores on a scale | 3.16 (0.63) | 3.46 (0.55) | 3.31 (0.63)

4. Secondary Outcome: Score of Visibility Assessment - Border Delineation by Blinded Reader
Description: Border delineation for each lesion on postcontrast MR images using the 4-point scale by averaged blinded reader (Score 1=None, 2=Moderate, 3=Good, 4=Excellent)
Time Frame: one day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 143 | 148 | 149
scores on a scale | 3.30 (0.46) | 3.45 (0.48) | 3.36 (0.56)

5. Secondary Outcome: Score of Visibility Assessment - Border Delineation by Investigator
Description: Border delineation for each lesion on postcontrast MR images using the 4-point scale by investigator (Score 1=None, 2=Moderate, 3=Good, 4=Excellent)
Time Frame: one day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 143 | 143 | 144
scores on a scale | 3.10 (0.70) | 3.38 (0.61) | 3.22 (0.68)

6. Secondary Outcome: Treatment Planning Confidence - Gadobutrol 0.1 mmol/kg bw vs. Gadoteridol (ProHance) 0.2 mmol/kg bw by Treatment Planning Experts (TPE)
Description: Treatment planning confidence evaluated separately for each image set (gadobutrol [Gado-] 0.1 mmol/kg bw and gadoteridol [Pro-] 0.2 mmol/kg) by TPE (category: not confident, confident, and not assessable)
Time Frame: one day
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Gadobutrol 0.1 mmol/kg bw vs. ProHance 0.2 mmol/kg bw: Participants with MR images after first injection of gadobutrol 0.1 mmol/kg bw (dose of 0.1 mmol/kg bw) and two injections of gadoteridol 0.1 mmol/kg bw (total dose of 0.2 mmol/kg bw)
Arm/Group | Gadobutrol 0.1 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 151
participants
  Gado-not confident, Pro-not confident | 0
  Gado-not confident, Pro-confident | 2
  Gado-not confident, Pro-not assessable | 0
  Gado-confident, Pro-not confident | 1
  Gado-confident, Pro-confident | 148
  Gado-confident, Pro-not assessable | 0
  Gado-not assessable, Pro-not confident | 0
  Gado-not assessable, Pro-confident | 0
  Gado-not assessable, Pro-not assessable | 0

7. Secondary Outcome: Treatment Planning Confidence - Gadobutrol 0.1 mmol/kg bw vs. Gadoteridol (ProHance) 0.2 mmol/kg bw by Investigator
Description: Treatment planning confidence evaluated separately for each image set (gadobutrol 0.1 mmol/kg bw and gadoteridol 0.2 mmol/kg) by investigator (category: not confident, confident, and not assessable)
Time Frame: one day
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Gadobutrol 0.1 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 151
participants
  Gado-not confident, Pro-not confident | 1
  Gado-not confident, Pro-confident | 0
  Gado-not confident, Pro-not assessable | 0
  Gado-confident, Pro-not confident | 0
  Gado-confident, Pro-confident | 149
  Gado-confident, Pro-not assessable | 0
  Gado-not assessable, Pro-not confident | 0
  Gado-not assessable, Pro-confident | 1
  Gado-not assessable, Pro-not assessable | 0

8. Secondary Outcome: Treatment Planning Confidence - Gadobutrol 0.2 mmol/kg bw vs. Gadoteridol (ProHance) 0.2 mmol/kg bw by TPE
Description: Treatment planning confidence evaluated separately for each image set (gadobutrol 0.2 mmol/kg bw and gadoteridol 0.2 mmol/kg) by TPE (category: not confident, confident, and not assessable)
Time Frame: one day
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Gadobutrol 0.2 mmol/kg bw vs. ProHance 0.2 mmol/kg bw: Participants with MR images after two injections of gadobutrol 0.1 mmol/kg bw (total dose of 0.2 mmol/kg bw) and two injections of gadoteridol 0.1 mmol/kg bw (total dose of 0.2 mmol/kg bw)
Arm/Group | Gadobutrol 0.2 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 151
participants
  Gado-not confident, Pro-not confident | 0
  Gado-not confident, Pro-confident | 1
  Gado-not confident, Pro-not assessable | 0
  Gado-confident, Pro-not confident | 0
  Gado-confident, Pro-confident | 150
  Gado-confident, Pro-not assessable | 0
  Gado-not assessable, Pro-not confident | 0
  Gado-not assessable, Pro-confident | 0
  Gado-not assessable, Pro-not assessable | 0

9. Secondary Outcome: Treatment Planning Confidence - Gadobutrol 0.2 mmol/kg bw vs. Gadoteridol (ProHance) 0.2 mmol/kg bw by Investigator
Description: Treatment planning confidence evaluated separately for each image set (gadobutrol 0.2 mmol/kg bw and gadoteridol 0.2 mmol/kg) by investigator (category: not confident, confident, and not assessable)
Time Frame: one day
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Gadobutrol 0.2 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 151
participants
  Gado-not confident, Pro-not confident | 1
  Gado-not confident, Pro-confident | 0
  Gado-not confident, Pro-not assessable | 0
  Gado-confident, Pro-not confident | 0
  Gado-confident, Pro-confident | 149
  Gado-confident, Pro-not assessable | 0
  Gado-not assessable, Pro-not confident | 0
  Gado-not assessable, Pro-confident | 1
  Gado-not assessable, Pro-not assessable | 0

10. Secondary Outcome: Number of Participants With Performance in Stereotactic Radiosurgery (SRS) Planning by TPE
Description: Comparison of overall image quality for SRS treatment planning between gadobutrol and gadoteridol by TPE
Time Frame: one day
Population: Participants without a major protocol deviation or conditions that could affect his or her efficacy evaluation (Per Protocol Set), whose images were assessed as "confident in treatment planning" with gadobutrol and ProHance, and who were assessed as applicable for SRS, and had valid data for this Outcome Measure
Measure: Number; unit: participants
Arm/Group | Gadobutrol 0.1 mmol/kg bw vs. ProHance 0.2 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 65 | 62
participants
  Gadobutrol was better than ProHance | 26 | 22
  ProHance was better than gadobutrol | 15 | 10
  Both image sets were comparable | 24 | 30

11. Secondary Outcome: Number of Participants With Performance in Stereotactic Radiosurgery (SRS) Planning by Investigator
Description: Comparison of overall image quality for SRS treatment planning between gadobutrol and gadoteridol by investigator
Time Frame: one day
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Gadobutrol 0.1 mmol/kg bw vs. ProHance 0.2 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 88 | 88
participants
  Gadobutrol was better than ProHance | 9 | 24
  ProHance was better than gadobutrol | 21 | 5
  Both image sets were comparable | 58 | 59

12. Secondary Outcome: Number of Participants With Reasons for Performance in SRS Planning by TPE
Description: Reasons for comparison results of overall image quality for SRS treatment planning between gadobutrol and gadoteridol by investigator (multiple answers applicable)
Time Frame: one day
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Gadobutrol 0.1 mmol/kg bw vs. ProHance 0.2 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 65 | 62
participants
  Gadobutrol was better: newly detected lesions | 2 | 5
  Gadobutrol was better: lesion size exceeds limit | 1 | 0
  Gadobutrol better: newly treatable lesions | 5 | 3
  Gadobutrol was better: extended radiation area | 8 | 5
  Gadobutrol was better: clarified radiation area | 15 | 11
  ProHance was better: newly detected lesions | 4 | 1
  ProHance was better: lesion size exceeds the limit | 1 | 0
  ProHance was better: newly treatable lesions | 4 | 2
  ProHance was better: extended radiation area | 3 | 5
  ProHance was better: clarified radiation area | 8 | 3

13. Secondary Outcome: Number of Participants With Reasons for Performance in SRS Planning by Investigator
Description: as for outcome 12
Time Frame: one day
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Gadobutrol 0.1 mmol/kg bw vs. ProHance 0.2 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw vs. ProHance 0.2 mmol/kg bw
Number analyzed (Participants) | 88 | 88
participants
  Gadobutrol better: newly treatable lesions | 2 | 8
  Gadobutrol was better: extended radiation area | 0 | 1
  Gadobutrol was better: clarified radiation area | 6 | 17
  Gadobutrol was better: other | 1 | 1
  ProHance was better: newly treatable lesions | 11 | 3
  ProHance was better: extended radiation area | 1 | 0
  ProHance was better: clarified radiation area | 8 | 2
  ProHance was better: other | 3 | 0

14. Secondary Outcome: Lesion Size Evaluated by Independent Radiologist
Description: Size of each lesion on postcontrast MR images evaluated by independent radiologist (mean and standard deviation of 603 lesions)
Time Frame: one day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 151 | 151 | 151
mm | 8.79 (8.06) | 9.07 (8.19) | 8.83 (8.02)

15. Secondary Outcome: Contrast Noise Ratio (CNR) of Lesions Evaluated by Independent Radiologist
Description: CNR of lesion/normal white matter based on the signal intensity of MR images evaluated by independent radiologist (mean and standard deviation of 306 lesions)
Time Frame: one day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CNR
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 151 | 151 | 151
CNR | 36.74 (47.82) | 60.09 (67.40) | 53.01 (56.20)

16. Secondary Outcome: Intraclass Correlation Coefficient (ICC) Among 3 Blinded Readers on the Number of Detected Lesions
Description: ICC among 3 blinded readers calculated for number of detected lesions using the statistical model with two random effects, i.e., blinded readers and individual patients.
Time Frame: one day
Population: as for outcome 1
Measure: Number; unit: ICC
Arm/Group | Gadobutrol 0.1 mmol/kg bw | Gadobutrol 0.2 mmol/kg bw | Gadoteridol (ProHance) 0.2mmol/kg bw
Number analyzed (Participants) | 151 | 151 | 151
ICC | 0.963 | 0.955 | 0.949

ADVERSE EVENTS:
Groups:
- Gadobutrol Period: Participants received two injections (i.v.) of gadobutrol 0.1 mmol/kg bw, corresponding to a total dose of 0.2 mmol/kg bw.
- ProHance Period: Participants received two injections (i.v.) of gadoteridol 0.1 mmol/kg bw, corresponding to a total dose of 0.2 mmol/kg bw.
Arm/Group | Gadobutrol Period | ProHance Period
Serious Adverse Events (participants affected / at risk) | 0/161 | 2/162
Other Adverse Events (participants affected / at risk) | 2/161 | 9/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol Period (N=161) | ProHance Period (N=162)
General physical health deterioration (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol Period (N=161) | ProHance Period (N=162)
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Glucose urine present (Investigations) | 0 | 2
Headache (Nervous system disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days